CLINICAL TRIAL: NCT03262870
Title: Gut Microbiota and Multiple Sclerosis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Azza Gama, Dr, Assiut University
Other Study IDs: GMAMS
Record Dates: First submitted 2017-08-24; First posted 2017-08-25 (Actual); Last update posted 2017-08-29 (Actual); Status verified 2017-08

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Gut microbiota and multiple sclerosis Multiple sclerosis is a pro-inflammatory demyelinating disease of the central nervous system.

DETAILED DESCRIPTION:
Multiple sclerosis is a pro-inflammatory demyelinating disease of the central nervous system. The etiology of MS is complex and poorly understood. Both genetic and environmental factors play a role and recent evidence suggests that gut microbiota is one of the key environmental factors. Gut microbiota is increasingly being seen an important environmental risk factor for multiple sclerosis, and strategies to correct an imbalance in intestinal flora.The first study, "Multiple sclerosis patients have a distinct gut microbiota compared to healthy controls," published in Scientific Reports, found that people with relapsing-remitting MS have altered fecal microbiota and may have microbial dysbiosis. People with MS had reduced levels of a protein called aryl hydrocarbon receptor circulating in their blood.Aryl hydrocarbon receptor is involved in many biological processes, including inflammation. The researchers found that gut microbiota play a role in turning tryptophan, and amino acid found in food, into Aryl hydrocarbon receptor agonists, which act on cells of the nervous system called astrocytes and limit inflammation of the central nervous system. Low levels of Aryl hydrocarbon receptor in multiple sclerosis patients may explain how microbial dysbiosis could be causing the condition.Increased constipation and fecal incontinence and increased gut permeability in multiple sclerosis patients, and increased occurrence of inflammatory bowel diseases in MS patients and their families suggest an important gut-central nevus system connection.Interestingly, gut bacteria can also influence the blood brain barrier integrity. These studiesimplicate that gut microbiota may potentially be operational in predisposition to or modification of the disease course of multiple sclerosis.

ELIGIBILITY:
Inclusion Criteria:

* The study will included 40 cases of MS according to Diagnostic criteria of multiple sclerosis they classified into two types of Multiple sclerosis ,Relapsing-remitting MS (group 1), and Primary progressive MS, Secondary progressive MS, and Progressive relapsing MS (group 2).

Each patient was submitted to the following:

Expanded disability status scale score between 1 and 6 and functional system score.

Demographic and clinical data (Age, sex, age of onset, severity of disease, clinical symptoms and signs, Types of treatment, duration of treatment, number of attacks).

Exclusion Criteria:

* The general exclusion criteria included prior surgeries, any patients or controls currently taking antibiotics or probiotic supplements,or having a known history of disease with an disease such, rheumatoid arthritis,type-1-diabetes, and IBD, were also excluded from the study.Microbial DNA was extracted from fecal material of each sample.

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients admitted in Assiut University hospital and outpatient clinic individuals
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2018-01-04 (Estimated); Primary Completion 2019-01-04 (Estimated); Study Completion 2020-01-04 (Estimated)

PRIMARY OUTCOMES:
Understanding the role of gut microbiota in the modification of the disease course of MS . | 24 month

IPD SHARING:
Plan to Share IPD: Undecided